CLINICAL TRIAL: NCT02974686
Title: Conversion From MPA to Zortress (Everolimus) for GI Toxicity Post-renal Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201603167; CRAD001AUS209T (Other Grant/Funding Number: Novartis Pharmaceuticals Company)
Record Dates: First submitted 2016-11-03; First posted 2016-11-28 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Kidney Transplant Rejection; Gastrointestinal Disorder, Functional
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (EVR) (Active Comparator): Patients experiencing gastrointestinal adverse effects in the first year post transplant will be converted from mycophenolate to everolimus
  Interventions: Drug: Everolimus
- Prior Agent (MPA) (Active Comparator): Patient will have baseline data collected while on MPA for comparison with EVR
  Interventions: Drug: Mycophenolic Acid

INTERVENTIONS:
Drug: Everolimus
  Other Names: Zortress
  Arms: Interventional (EVR)
Drug: Mycophenolic Acid
  Other Names: Cellcept; Myfortic
  Arms: Prior Agent (MPA)

SUMMARY:
Patients who receive renal transplantation at Barnes Jewish Hospital (BJH) are placed on triple maintenance immunosuppression, which means that patients take 3 types of immunosuppression drugs to suppress their immune system including tacrolimus, mycophenolate (MPA), and prednisone. However, due to the effects of MPA on the gastrointestinal tract, patients often complain of GI adverse effects. Current practice is to either dose-reduce MPA or convert the patient to an alternative agent, typically Azathioprine. Both of these strategies have limitations, largely due to concerns related to efficacy. Everolimus (EVR) has demonstrated similar efficacy to MPA in renal transplantation and may offer a benefit related to GI adverse effects, so the investigators will convert patients to EVR in this study. Patients who are within their first year post-transplant will be converted to EVR upon enrollment in the study, and serial measurements ,or a series of measurements looking for an increase or decrease over time, of GI adverse effects will be conducted over 1 year post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipients at Washington University/Barnes-Jewish Hospital
2. Experiencing GI toxicity from MPA as determined by the treating physician within 12 months post-renal transplant
3. On standard immunosuppression with tacrolimus and prednisone

Exclusion Criteria:

1. Dual organ or kidney after another solid organ transplant
2. Presence of a preexisting significant GI condition that does not have a presumed causal relationship with MPA
3. Evidence of any GI disorder induced by an infection, underlying medical condition, or concomitant medication other than MPA
4. Estimated glomerular filtration rate (eGFR) <40 ml/min at time of possible conversion
5. Proteinuria >1 gram/day at time of possible conversion
6. Profound bone marrow suppression at the time of possible conversion as defined as:

   * Hemoglobin <10 g/dL
   * White blood cell (WBC) < 3 K/cumm
   * Platelets <100 K/cumm
7. Wound healing issues at time of possible conversion (eg, wound dehiscence, wound infection, incisional hernia, lymphocele, seroma)
8. Elevated total cholesterol (>350 mg/dL) and/or triglycerides (>500 ng/dL) at time of possible conversion
9. Hypersensitivity to everolimus, sirolimus, or other rapamycin derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Groups:
- Interventional Everolimus (EVR): Patients experiencing gastrointestinal adverse effects in the first year post transplant will be converted from mycophenolate to everolimus
  Everolimus
- Prior Agent Mycophenolic Acid (MPA): Patient will have baseline data collected while on MPA for comparison with EVR
  Mycophenolic Acid
Period: Overall Study
Arm/Group | Interventional Everolimus (EVR) | Prior Agent Mycophenolic Acid (MPA)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Groups:
- Interventional (EVR): Patients experiencing gastrointestinal adverse effects in the first year post transplant will be converted from mycophenolate to everolimus
  Everolimus
- Prior Agent (MPA): Patient will have baseline data collected while on MPA for comparison with EVR
  Mycophenolic Acid
- Total: Total of all reporting groups
Arm/Group | Interventional (EVR) | Prior Agent (MPA) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Symptom Rating Scale
Description: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Time Frame: 3 months
Population: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Arm/Group | Interventional (EVR) | Prior Agent (MPA)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Gastrointestinal Symptom Rating Scale
Description: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Time Frame: 1, 6, and 12 months
Population: Trial was terminated with only 1 participant enrolled, no data is reported to protect patient confidentiality
Arm/Group | Interventional (EVR) | Prior Agent (MPA)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Biopsy Proven Acute Rejection
Description: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Time Frame: 12 months
Population: Trial was terminated with only 1 participant enrolled, no data is reported to protect patient confidentiality
Arm/Group | Interventional Everolimus (EVR) | Prior Agent Mycophenolic Acid (MPA)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Description: Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.
Arm/Group | Interventional (EVR) | Prior Agent (MPA)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Trial was terminated with only 1 participant enrolled. No data is reported here to maintain patient confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT02974686/Prot_SAP_000.pdf